CLINICAL TRIAL: NCT07305818
Title: A Phase 1 First-in-Human, Single and Multiple Ascending Dose Study to Evaluate Safety Tolerability Pharmacokinetics Pharmacodynamics, and Immunogenicity of Intravenous and Subcutaneous Administration of MER511 in Adults With Graves' Disease
Brief Title: NEXUS Study: A Study to Test Single and Multiple Doses of MER511 Given to Adults With Graves' Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merida Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MER511-1001; 2025-523823-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Graves Disease
Keywords: Graves' Disease; Hyperthyroidism; Basedow disease; Exophthalmic goitre; TSHR; Autoimmune; Anti-thyroid drugs; Autoimmune thyroid disease
MeSH Terms: conditions — Graves Disease; Hyperthyroidism

STUDY DESIGN:
Intervention Model Description: The study will enroll cohorts of participants who will be assigned to a dose group for Part A and Part B.
Who Masked: Participant, Investigator
Masking Description: Sponsor-open label, participant- and investigator-blind (Masked)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (SAD) MER511 IV (Experimental): For Cohorts 1-7 , each cohort participant will receive a single ascending dose of MER511 via IV administration on Day 1
  Interventions: Biological: MER511 (IV)
- Part A (SAD) placebo IV (Placebo Comparator): For Cohorts 1-7, each cohort participant will receive a single dose of placebo via IV administration on Day 1
  Interventions: Biological: Placebo comparator (IV)
- Part A (SAD) MER511 SC (Experimental): For Cohort 8, participants will receive a single dose of MER511 (determined from Cohort 1-7) via SC administration on Day 1
  Interventions: Biological: MER511 (SC)
- Part A (SAD) placebo SC (Placebo Comparator): For Cohort 8, participants will receive a single dose of placebo (determined from Cohort 1-7) via SC administration on Day 1
  Interventions: Biological: Placebo comparator (SC)
- Part B (MAD) MER511 SC (Experimental): Up to 3 cohorts of participants will receive multiple ascending doses of MER511 via SC administration assigned for their cohort on Day 1 and Day 29
  Interventions: Biological: MER511 (SC) for MAD
- - Part B (MAD) placebo SC (Placebo Comparator): Up to 3 cohorts of participants will receive multiple doses of placebo via SC administration assigned for their cohort on Day 1 and Day 29
  Interventions: Biological: Placebo comparator (SC) for MAD

INTERVENTIONS:
Biological: MER511 (IV) — Participants will receive a single dose of MER511 on Day 1
  Arms: Part A (SAD) MER511 IV
Biological: Placebo comparator (IV) — Participants will receive a single dose of Placebo on Day 1
  Arms: Part A (SAD) placebo IV
Biological: MER511 (SC) — Participants will receive a single dose of MER511 on Day 1
  Arms: Part A (SAD) MER511 SC
Biological: Placebo comparator (SC) — Participants will receive a single dose of Placebo on Day 1
  Arms: Part A (SAD) placebo SC
Biological: MER511 (SC) for MAD — Participants will receive multiple ascending doses of MER511 via SC administration assigned for their cohort on Day 1 and Day 29
  Arms: Part B (MAD) MER511 SC
Biological: Placebo comparator (SC) for MAD — Participants will receive multiple doses of placebo via SC administration assigned for their cohort on Day 1 and Day 29
  Arms: - Part B (MAD) placebo SC

SUMMARY:
The purpose of this study is to evaluate how well MER511 is tolerated and what side effects may occur in adults who have Graves' disease. The study drug will be administered either intravenously (into a vein in the arm) or subcutaneously (under the skin).

Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body.

DETAILED DESCRIPTION:
This Phase 1, first-in-human, multicenter study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of single and multiple ascending doses of MER511 administered to adults (18 to 55 years of age, inclusive) with GD (Graves' disease).

The study will consist of 2 sequential parts: a single ascending dose (SAD) part (Part A) followed by a multiple ascending dose (MAD) part (Part B).

Part A will employ a placebo-controlled, sponsor-open, participant- and investigator-blind design to evaluate the safety, tolerability, PK, PD, and immunogenicity of single ascending intravenous doses and a single subcutaneous dose of MER511.

Part B will employ a placebo-controlled, sponsor-open, participant- and investigator-blind design to assess the safety, tolerability, PK, PD, and immunogenicity of multiple subcutaneous doses of MER511.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 55 years of age, inclusive, at the time of signing the ICF
2. Documented GD diagnosis,
3. Receiving stable dose of ATD (Antithyroid drug)
4. Body weight at least 50 kg (110 lb) and body mass index (BMI) 18.0-35.0 kg/m2, inclusive
5. Women of childbearing potential must agree to use highly effective contraceptive methods
6. Men with partners of childbearing potential or who are pregnant must agree to use a condom or strict abstinence
7. Signed informed consent to participate in the study
8. Willingness and ability, in the opinion of the investigator, to comply with protocol requirements and restrictions (eg, dosing, schedule of assessments).

Exclusion Criteria:

1. History of:

   1. total thyroidectomy.
   2. History of hyperthyroidism not caused by GD (eg, toxic adenoma, toxic multinodular goiter).
   3. History of thyroid storm.
   4. History of agranulocytosis, anemia, leukopenia, thrombocytopenia, vasculitis, or liver toxicity due to prior ATD therapy Treatment with RAI therapy within 12 months prior to Screening
2. Likely to require definitive treatment for GD (RAI therapy or thyroidectomy) during the study, based on GD history and anticipated prognosis.
3. Use of levothyroxine, desiccated thyroid extract, or T3 at any dose within 6 weeks prior to Screening.
4. History of active or chronic moderate-to-severe TED per EUropean Group On Graves' Orbitopathy (EUGOGO) criteria as judged by the investigator at Screening
5. History of TED-directed medical treatment (including IV/oral steroids, immunosuppressants, or teprotumumab), surgical treatment, and/or orbital radiation.
6. Major surgery or use of iodinated contrast within 3 months prior to planned IMP dosing.
7. Active systemic autoimmune disease requiring treatment that causes undue risk in the opinion of the investigator.
8. History of cardiovascular, respiratory, renal, gastrointestinal, endocrinological (other than GD), hematological, immunodeficiency, or neurological disorders that may constitute a risk when taking the IMP or interfere with data interpretation.
9. History of liver disease
10. Pregnant, breastfeeding, or planning to become pregnant during the study
11. Treatment with prohibited medications prior to planned IMP dosing or likely to require prohibited concomitant therapy during the study
12. Live vaccine(s) or mRNA vaccine(s) within 1 month prior to IMP dosing, or plans to receive such vaccines during the study
13. Treatment with any investigational drug within 6 months prior to enrollment
14. Total IgG level <700 mg/dL at Screening
15. Any of the following at Screening (confirmed by single repeat measurement, if deemed necessary):

    * ALT or AST >1.5 × ULN
    * Total bilirubin >1.5 × ULN
16. Estimated glomerular filtration rate (eGFR) <85 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation
17. Positive result for HIV antibody, HBsAg, or hepatitis C antibody with detectable viral RNA levels at Screening
18. Positive drug screen or positive test for alcohol
19. 12-lead ECG demonstrating any of the following at Screening:

    * QTcF interval >450 ms
    * QRS interval >120 ms
    * PR interval >220 ms
20. 20. Blood pressure measurements demonstrating any of the following at Screening:

    * Systolic blood pressure ≥140 mmHg
    * Diastolic blood pressure ≥90 mmHg
21. Heart rate <45 bpm or >100 bpm
22. Donated more than 500 mL of blood in the 2 months prior to signing the ICF
23. Current enrollment or past participation within 30 days or 5 half-lives (whichever is longer) prior to signing the ICF in any other clinical trial involving an IMP
24. Refusal to adhere to lifestyle considerations as defined in the protocol
25. Employee of the investigator, clinic, or sponsor with direct involvement in the proposed study or other studies under the direction of the investigator or clinic, as well as family members of the employee or investigator
26. Any other conditions that, in the opinion of the investigator or the sponsor, could interfere with participation in or completion of the study
27. Part B only: anyone who received IMP during Part A of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2028-07-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with TEAEs (Treatment-emergent adverse events) | - Part A (SAD) Cohorts: Day 1 up to Week 16 - Part B (MAD) Cohorts: Day 1 up to Week 24
  Adverse events that start or worsen in severity after the start of study drug will be categorized as TEAEs
Number of participants with clinically significant changes in ECGs, vital signs, clinical laboratory values, and physical examination | - Part A (SAD) Cohorts: Day 1 up to Week 16 - Part B (MAD) Cohorts: Day 1 up to Week 24
  Incidence of clinically significant abnormalities in ECGs, vital signs, clinical laboratory values, and physical examination

SECONDARY OUTCOMES:
Serum Cmax (Maximum observed concentration) | - Part A (SAD) Cohorts: Day 1 (Week 0 dosing day) through Week 16- Part B (MAD) Cohorts: Day 1 (Week 0 dosing Day) Through Week 24
  Measurement of the maximum observed concentration
Serum tmax (Time to maximum concentration) | - Part A (SAD) Cohorts: Day 1 (Week 0 dosing day) Through Week 16 - Part B (MAD) Cohorts: Day 1 (Week 0 dosing day) Through Week 24
  Measurement of the time to maximum observed concentration
Serum AUCinf (area under concentration-time curve from time zero to infinity) | Part A (SAD) Only: Day 1 (Week 0) Dosing Through Week 16
  Measurement of area under concentration-time curve from time zero to infinity
Serum AUC0-tau (area under concentration-time curve during the dosing interval) | Part B (MAD) Only: Day 1 (Week 0) Dosing Through Week 24
  Measurement of area under concentration-time curve during the dosing interval
Number of participants with ADAs (Anti-drug antibody) | - Part A (SAD) Cohorts: Day 1 (Week 0) Dosing Through Week 16 or Early Discontinuation - Part B (MAD) Cohorts: Day 1 (Week 0) Dosing Through Week 24
  Blood samples will be collected to evaluate the immunogenicity of MER511 in participants with GD (Graves' disease)

CONTACTS AND LOCATIONS:
Locations (1):
- Site # 1101, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No